CLINICAL TRIAL: NCT00030784
Title: Phase I Study To Determine The Safety Of Caelyx (Doxorubin HCI, Pegylated Liposomal) In Combination With Ifosfamide In Previously Untreated Adult Patients With Advanced And/Or Metastatic Soft Tissues Sarcomas
Brief Title: Liposomal Doxorubicin Plus Ifosfamide in Treating Patients With Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-62002; EORTC-62002
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; stage III adult soft tissue sarcoma; adult alveolar soft-part sarcoma; adult epithelioid sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult rhabdomyosarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Sarcoma, Alveolar Soft Part; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Rhabdomyosarcoma | interventions — Ifosfamide

INTERVENTIONS:
Drug: ifosfamide
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining liposomal doxorubicin with ifosfamide in treating patients who have advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of ifosfamide in combination with doxorubicin HCl liposome in patients with previously untreated advanced or metastatic soft tissue sarcoma.
* Determine the objective response in patients treated with this regimen.
* Determine the dose-limiting toxicity in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of ifosfamide.

Patients receive doxorubicin HCl liposome IV over 1 hour on day 1 and ifosfamide IV over 4 hours on days 1-3 OR on days 1-4 (for patients enrolled on dose level 6). Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ifosfamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 8 weeks until disease progression and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma

  * Advanced and/or metastatic disease
  * Must be of any of the following types:

    * Malignant fibrous histiocytoma
    * Liposarcoma (excluding lipomas and well-differentiated liposarcomas)
    * Rhabdomyosarcoma
    * Synovial sarcoma
    * Malignant paraganglioma
    * Fibrosarcoma
    * Leiomyosarcoma
    * Angiosarcoma
    * Neurogenic sarcoma
    * Sarcoma not otherwise specified
  * Paraffin blocks and slides must be available
* Measurable disease

  * Osseous lesions and pleural effusions are not considered measurable disease
* Evidence of progressive disease within the past 6 weeks
* The following conditions are excluded:

  * Gastrointestinal stromal tumors
  * Malignant mesothelioma
  * Chondrosarcoma
  * Neuroblastoma
  * Osteosarcoma
  * Ewing's sarcoma
  * Embryonal rhabdomyosarcoma
* No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.75 mg/dL
* Albumin at least 2.5 g/dL

Renal:

* Creatinine no greater than 1.4 mg/dL
* Creatinine clearance at least 65 mL/min

Cardiovascular:

* Ejection fraction at least 50% by echocardiogram or isotopic methods
* No history of cardiovascular disease

Other:

* No other prior or concurrent primary malignancies except adequately treated carcinoma in situ of the cervix or basal cell carcinoma
* No other severe medical illness
* No psychosis
* No psychological, familial, sociological, or geographical condition that would preclude study participation
* Not pregnant
* Fertile patients must use effective contraception (barrier method for men) during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for advanced disease
* No other concurrent systemic chemotherapy for malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to sole indicator lesion
* Concurrent radiotherapy allowed except to sole indicator lesion

Surgery:

* Not specified

Other:

* No other concurrent investigational drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-11; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ole S. Nielsen, MD, Study Chair — Aarhus Universitetshospital - Aarhus Sygehus
Locations (2):
- Aarhus University Hospital - Aarhus Sygehus - Norrebrogade, Aarhus, Denmark
- Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin, Germany